CLINICAL TRIAL: NCT03635814
Title: Multi-center, Randomized, Double-blind, Dose-finding, Phase 2a Clinical Trial to Evaluate the Effecacy and Safety of YD312 Tablet in Patients With Diabetic Macular Edema
Brief Title: The Study to YD312 Tablet in Patients With Diabetic Macular Edema
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: YD Global Life Science Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YD312-01-P2
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Macular Edema(DME)
Keywords: Clinicaltrial, DME, DR, AMD, imatinib mesylate

STUDY DESIGN:
Intervention Model Description: Subjects who finally meet inclusion/exclusion criteria will be randomized into lower dose group (YD312 Tablet 50 mg), middle dose group (YD312 Tablet 150 mg), higher dose group (YD312 Tablet 350 mg), and placebo group as a ratio of 1:1:1:1 and the relevant investigational product will be administered for 12 weeks.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- YD312 drug treatment (Experimental): From the date when dispensed, investigational products will be dosed once a day at similar time to the first dosing time with meals and much water.
  Interventions: Drug: YD312 50mg; Drug: YD312 150mg; Drug: YD312 350mg
- YD312 placebo drug treatment (Placebo Comparator): From the date when dispensed, investigational products will be dosed once a day at similar time to the first dosing time with meals and much water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YD312 50mg — YD312 50mg * 1 + placebo 6 tablets
  Arms: YD312 drug treatment
Drug: YD312 150mg — YD312 50mg * 3 + placebo 6 tablets
  Arms: YD312 drug treatment
Drug: YD312 350mg — YD312 50mg * 7 tablets
  Arms: YD312 drug treatment
Drug: Placebo — YD312 0mg * 7 tabets
  Arms: YD312 placebo drug treatment

SUMMARY:
This study objectives is to evaluate the efficacy of YD312 to improve visual acuity in patients with diabetic macular edema (DME) compared to placebo and determine optimal dose of phase 2b study.

DETAILED DESCRIPTION:
These study results present the possibility that imatinib can be used as a new DME inhibiting agent by involving VEGF-independent ocular angiogenesis, not action points of existing agents, in effectively inhibiting excessive vascular angiogenesis observed in oxygen-induced retinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Screening Inclusion Criteria

   Study subjects must be eligible for the following criteria at screening:
   1. Subject who is male or female ≥ 19 years of age
   2. Subject who has a diagnosis of Type 1 or 2 diabetes
   3. Subject who has study eye with definite retinal thickening due to diabetic macular edema involving the center of the macula
   4. Subject who has voluntarily signed an informed consent form
2. Randomization Inclusion Criteria

Study eye must be eligible for the following criteria at randomization:

1. Subject who has study eye with central subfield thickness (CST) of ≥ 300 μm on optical coherence tomography (OCT)
2. Subject who has study eye with an early treatment diabetic retinopathy study (ETDRS) best-corrected visual acuity (BCVA) letter score ranging from 39 to 78, inclusive (approximate Snellen equivalent of 20/32 - 20/160)

Exclusion Criteria:

1. Subject who has study eye with any of the following criteria:

   1. Subject whose primary cause of macular edema is non-diabetic disease/condition (e.g., cataract extraction, vitreomacular interface abnormalities)
   2. Subject who is expected to have no improvement of decreased visual acuity in the opinion of investigator, even if macular edema is resolved (e.g., foveal atrophy, abnormal pigmentation, dense subfoveal hard exudate)
   3. Subject who has proliferative diabetic retinopathy.
   4. Subject who took the following within 3 months before randomization

      ① Focal/grid laser photocoagulation

      ② Intravitreal/circumbulbar corticosteroid, anti-VEGF and pro-VEGF (but, no wash-out period is required for the corticosteroid eyedrops)
   5. Subject who took panretinal photocoagulation (PRP) or intravitreal dexamethasone implant within 6 months before randomization
   6. Subject who has a history of vitrectomy
   7. Subject who took major ophthalmic surgeries (all intraocular surgeries including cataract extraction and scleral buckle) within 6 months before randomization
2. Subject who had systemic treatment of corticosteroid or anti-VEGF within 3 months before randomization.
3. Subject who administered vaccinium myrtillus extract or dobesilate calcium within 2 weeks before randomization
4. Subject who is suspected to require administration/treatment of drug/procedure that may affect the efficacy evaluation before the participation of clinical trial or during clinical trial (refer to '10.4 Combination Therapy and Contraindication').
5. Subject who has the following illness or abnormal laboratory test values:

   1. Subject who has a hypersensitivity to any excipients of the investigational product or similar class of drug and ingredient
   2. Subject who has uncontrolled hypertension (SBP > 160 mmHg or DBP >100 mmHg)
   3. Subject who has uncontrolled diabetes (HbA1c > 10.0%)
   4. Subject who has uncontrolled glaucoma in either eye (intraocular pressure (IOP) > 24 mmHg on medication or according to the investigator's judgment)
   5. ANC < 1.5 × 109/L
   6. Platelet < 125 × 109/L
   7. Total bilirubin > 1.5 × ULN
   8. AST or ALT > 2 × ULN
   9. Clcr* < 40 mL/min

      * Clcr (Cockcroft-Gault formula)

      = [(140 - age) x weight(kg) (x 0.85 for females)] / [72 x serum creatinine (Scr) (mg/dL)]
   10. Severe heart failure (NYHA class III/IV)
   11. Malignant tumor within 5 years before randomization
   12. Subject who is known to be HIV positive, is active hepatitis B patient or carrier, or is hepatitis C patient
   13. Ocular inflammatory diseases such as uveitis, conjunctivitis, and blepharitis in either eye. However, the participation of subject in this study is considered at the discretion of investigator.
   14. Unstable angina, myocardial infarction, transient ischemic attack, cerebral infarction, coronary artery bypass surgery, or transluminal coronary angioplasty within 6 months before screening
6. Pregnant woman, lactating woman, or female or male subject of childbearing potential

   *hormonal contraceptives, intrauterne contraceptive device, sterilization of spouse (e.g., vasectomy, tubal ligation), double-barrier method (e.g., combinational use of spermicides and condoms, diaphragm, contraceptive sponge, of FemCap)
7. Subject who took administraion/procedure of other investigational products or medical devices within longer period between 30 days before screening or over 5time half-life.
8. Subject, at the discretion of the investigator, who is unsuitable to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in ETDRS BCVA latter score from baseline at Week 12 ( ETDRS chart reading at least 3 letters) | BCVA ERDRS measure at V1(screening), V2(baseline,week0), V3(week4), V4(week8), V5(week12)

SECONDARY OUTCOMES:
Change in ETDRS BCVA latter score from baseline at Weeks 4 and 8 | BCVA ERDRS measure at V1(screening), V2(baseline,week0), V3(week4), V4(week8), V5(week12)
Improvement or worsening rate of ETDRS BCVA from baseline at Weeks 4, 8, and 12 | BCVA ERDRS measure at V1(screening), V2(baseline,week0), V3(week4), V4(week8), V5(week12)
  * Proportion of improved subjects: ≥ 1 letter score increase, ≥ 10 letter score increase, ≥ 15 letter score increase
  * Proportion of worsened subjects: ≥ 5 letter score decrease, ≥ 10 letter score decrease, ≥ 15 letter score decrease
Change in CST from baseline at Weeks 4, 8, and 12 | BCVA ERDRS measure at V1(screening), V2(baseline,week0), V3(week4), V4(week8), V5(week12)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (13):
  - AXIS Clinical Trials, Los Angeles, California
  - South Flolida Clinical Trials, Hialeah, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Retina Associates, Chicago, Illinois
  - Elman Retina Group, Baltimore, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Impact Clinical Trials LV, Las Vegas, Nevada
  - NY Clinical Trials, New York, New York
  - Vitro-Retinal Consultants, Inc, Painesville, Ohio
  - Phensylvania Retina Specialists, Camp Hill, Pennsylvania
  - WR-Clinsearch, LLC, Chattanooga, Tennessee
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Wagner Macula & Retina Center, Norfolk, Virginia
- South Korea (7):
  - Kyungpook National University Hospital, Daegu, Chung-gu
  - Chungnam National University Hospital, Daejeon, Chung-gu
  - Samsung Medical Center, Seoul, Gangmam-gu
  - Kangnam Severance Hospital, Seoul, Gangnam-gu
  - Inje National University Busan Park Hospital, Busan, Jin-gu
  - Hanyang University Guri Medical Center, Guri-si, Kyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Kyeonggi-do

IPD SHARING:
Plan to Share IPD: Undecided